CLINICAL TRIAL: NCT01818609
Title: Influence of Reduce Daily Step Count on Muscle Protein Metabolism in Older Persons
Brief Title: Study of Inactivity on Metabolism of Elderly Muscles
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 267
Record Dates: First submitted 2011-07-19; First posted 2013-03-26 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2013-03

CONDITIONS: Sarcopenia
Keywords: sarcopenia; muscle; reduced activity; insulin sensitivity; protein; step reduction; muscle protein synthesis; whey protein; leg strength; whole body protein
MeSH Terms: conditions — Sarcopenia; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Step Reduction (Experimental): Step reduction:
  * Take less than 1500 steps/d
  * No disease
  Interventions: Behavioral: Step reduction

INTERVENTIONS:
Behavioral: Step reduction — taking less than 1500 steps/d
  Other Names: Sedentary behaviour

SUMMARY:
Skeletal muscle mass declines with inactivity (casting is a good example) and increases with activity (such as weightlifting). Whether muscle mass increases or decreases, is determined by whether more new proteins within muscle are made than are broken down. The investigators know that feeding protein increases the synthesis of new proteins but that the response of older muscles to protein feeding is blunted compared with the young. This resistance of the elderly to muscle building stimuli may be the primary reason that muscle mass is lost in aging. The investigators also know that periods of muscle disuse such as casting result in a person's muscle shrinking due, the investigators believe, to a lower rate of synthesis of new muscle proteins. Age-related muscle loss begins around 50 years old and proceeds at approximately 1% for every year after. Elderly persons would likely fare well with advancing age if their muscle loss were simply linear; however, a rate of muscle loss of 1% annually is a 'population view' and does not represent what occurs during short periods of muscle disuse (i.e. during hospitalization or illness), which occur with increasing frequency in elderly persons. During periods of disuse, the resistance of elderly muscles to protein nutrition may be worsened. The investigators will measure how quickly new proteins are made at rest and after protein feeding in elderly men, before and after a 14 day period of reduced activity brought on by having people reduce their daily step count.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Aged 60 to 80 years old
* Non-smoker Generally healthy and can tolerate the resistance exercise and protein drink

Exclusion Criteria:

* Allergies to whey protein
* Health problems such as: heart disease, rheumatoid arthritis of the knee joint, diabetes, poor lung function, uncontrolled hypertension, or any health conditions that might put participants at risks for this study
* Failed an exercise stress test
* Taking metformin and/or other medications for the control of blood glucose even though one might not be classified as diabetic
* Taking prescribed blood thinners such as warfarin and heparin but excluding aspirin
* Taking medications for lung and kidney conditions but excluding medication for asthma that is under control

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Fractional synthetic rate (FSR) of myofibrillar muscle protein | over 5h
  rate of making new muscle proteins

SECONDARY OUTCOMES:
Blood amino acid concentrations | over 5h
  concentration of amino acids in blood
Intramuscular signalling protein status | over 5h
  phosphorylation of key signalling proteins
Insulin sensitivity via blood sampling | over 5h
  measure of insulin concentration

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Phillips, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada